CLINICAL TRIAL: NCT00153842
Title: Phase I and II Clinical Studies of Paclitaxel and Carboplatin in Combination With Bexarotene Oral Capsules for the Treatment of Patients With Advanced Non-Small Cell Lung Cancer
Brief Title: A Study of Paclitaxel and Carboplatin in Combination With Bexarotene Oral Capsules in Patients With Advanced Lung Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: other trials show no survival benefit of bexarotene with platinum-based chemo
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: Bristol-Myers Squibb (Industry); Ligand Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D-0109
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Results first posted 2019-03-06 (Actual); Last update posted 2019-03-06 (Actual); Status verified 2019-02

CONDITIONS: Carcinoma, Non-small-cell Lung
Keywords: NSCLC; Bexarotene; Targretin
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Bexarotene

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bexarotene (Experimental): Bexarotene oral capsules will be administered daily beginning on the initial day of chemotherapy (day 1).
  Interventions: Drug: Bexarotene (targretin)

INTERVENTIONS:
Drug: Bexarotene (targretin) — Bexarotene oral capsules will be administered daily beginning on the initial day of chemotherapy (day 1).
  Level 1: 300 mg
  Other Names: Targretin, LGD1069
Drug: Bexarotene (targretin) — Bexarotene oral capsules will be administered daily beginning on the intitial day of chemotherapy (Day 1).
  Level 2: 400 mg
  Other Names: Targretin, LGD1069

SUMMARY:
The primary aim is to evaluate the safety (Phase I components) of administering bexarotene (Targretin®, LGD1069) oral capsules in combination with two Taxol® and carboplatin (Paraplatin®) schedules to patients with stage IIIB and IV non-small cell lung cancer. This study will also evaluate the preliminary efficacy (Phase II component) of bexarotene oral capsules in combination with the weekly Taxol® schedule and carboplatin in these patients.

DETAILED DESCRIPTION:
The phase I portion of the study will evaluate the safety of administering bexarotene oral capsules daily at two dose levels (300 mg/m2 and 400 mg/m2) in combination with carboplatin and Taxol®. At least 6 patients will be entered onto each dose level. Doses will not be escalated over the course of treatment of an individual patient. The recommended Phase II dose is defined as the highest dose of bexarotene oral capsules (300 mg/m2 or 400 mg/m2) in combination with carboplatin and Taxol® that induces DLT in fewer than or equal to 33% of patients.

The sequential phase II portion of the study will evaluate the efficacy of bexarotene oral capsules in combination with carboplatin and weekly Taxol® in patients with advanced non-small cell lung cancer. The efficacy will be gauged according to the rate of major response where, by definition, a major response occurs if a patient achieves either complete remission (CR) or partial remission (PR). For these patients a true response rate of 20% or greater is sufficiently large to warrant further investigation. A true response rate of 10% or less indicates that the combination is less active.

ELIGIBILITY:
Inclusion Criteria:

* unresectable stage IIIB or IV NSCLC
* adequate bone marrow, hepatic, thyroid and renal function

Exclusion Criteria:

* peripheral neuropathy >= grade 2
* gastrointestinal abnormalities
* known hypersensitivity to retinoids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2001-08; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James R Rigas, MD, Principal Investigator — Norris Cotton Cancer Center
Locations (1):
- Norris Cotton Cancer Center, Lebanon, New Hampshire, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase IB: Bexarotene 300mg vs 400mg administered with paclitaxel and carboplatin
- Phase II: Bexarotene 400mg in combination with Paraplatin and weekly Taxol.
Period: Overall Study
Arm/Group | Phase IB | Phase II
Started | 26 | 7
Completed | 26 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase IB | Phase II | Total
Number analyzed (Participants) | 26 | 7 | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 19 | 6 | 25
  >=65 years | 7 | 1 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.35 (9.79) | 57 (13.99) | 58.85 (10.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 2 | 13
  Male | 15 | 5 | 20
Region of Enrollment [Number; unit: participants]
  United States | 26 | 7 | 33

OUTCOME MEASURES:

1. Primary Outcome: Bexarotene Oral Capsules Safety at Two Dose Levels (300 mg/m2 and 400 mg/m2) in Combination With Carboplatin and Taxol®.
Description: At least 6 patients will be entered onto each dose level. Doses will not be escalated over the course of treatment of an individual patient. For the purpose of this protocol, an initial-dose-limiting toxicity (IDLT) is defined as a clinical observation that is, in the judgment of the Investigator, both attributable to the administration of bexarotene and necessitates a reduction in dose, suspension or discontinuation of study drug because of a NCI CTC Grade 3 or 4 level toxicity (with the exception of elevated lipids).
Time Frame: 36 months
Measure: Number; unit: participants experiencing IDLT
Groups:
- Phase IB: Bexarotene 300mg, Paclitaxel and Carboplatin: Bexarotene 300mg administered with paclitaxel and carboplatin
- Phase IB: Bexarotene 400mg, Paclitaxel and Carboplatin: Bexarotene 400mg administered with paclitaxel and carboplatin
- Phase II: Bexarotene 400mg administered with paclitaxel and carboplatin (Paraplatin and weekly Taxol)
Arm/Group | Phase IB: Bexarotene 300mg, Paclitaxel and Carboplatin | Phase IB: Bexarotene 400mg, Paclitaxel and Carboplatin | Phase II
Number analyzed (Participants) | 14 | 12 | 7
participants experiencing IDLT | 1 | 1 | 0

ADVERSE EVENTS:
Groups:
- Phase IB - Bexarotene 300mg, Paclitaxel and Carboplatin: Bexarotene 300mg administered with paclitaxel and carboplatin
- Phase IB - Bexarotene 400mg, Paclitaxel and Carboplatin: Bexarotene 400mg administered with paclitaxel and carboplatin
Arm/Group | Phase IB - Bexarotene 300mg, Paclitaxel and Carboplatin | Phase IB - Bexarotene 400mg, Paclitaxel and Carboplatin | Phase II
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/12 | 0/7
Serious Adverse Events (participants affected / at risk) | 1/14 | 0/12 | 2/7
Other Adverse Events (participants affected / at risk) | 0/14 | 0/12 | 0/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase IB - Bexarotene 300mg, Paclitaxel and Carboplatin (N=14) | Phase IB - Bexarotene 400mg, Paclitaxel and Carboplatin (N=12) | Phase II (N=7)
Myelosuppression (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertriglyceridemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes